CLINICAL TRIAL: NCT04622384
Title: The Performance of Renal Doppler Ultrasound in Predicting Outcome of Dialysis Weaning
Status: Completed | Type: Observational
Sponsor: Johan Fridolf Hermansen (Other)
Responsible Party: Sponsor-Investigator, Johan Fridolf Hermansen, Principal Investigator, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: 1-10-72-40-20(3)
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Acute Kidney Injury; Acute Kidney Failure Stage 3
Keywords: Ultrasound; Renal Replacement Therapy; Dialysis; Renal Doppler Ultrasound
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU patients: Patients who are treated with dialysis as CRRT and planned to undergo dialysis weaning.
  Interventions: Other: Dialysis weaning

INTERVENTIONS:
Other: Dialysis weaning — Dialysis weaning as planned by the attending ICU-physician.

SUMMARY:
Acute kidney injury (AKI) is a frequent problem in the intensive care unit (ICU) affecting more than 50 % of patients. AKI is associated with several adverse outcomes, including increased mortality and increased length of ICU- and hospital stay, in particular in patients requiring Renal Replacement Therapy (RRT).

Choosing the optimal time for attempting liberation from RRT is still unclear. With this study, we will describe the ability of renal ultrasound in predicting the outcome of dialysis weaning.

ELIGIBILITY:
Inclusion Criteria:

* All patients ≥ 18 years admitted to the ICU, Aarhus University Hospital who are treated with dialysis as continuous renal placement therapy (CRRT) and planned to undergo dialysis weaning

Exclusion Criteria:

* Insufficient ultrasonographic imaging of the kidneys
* Known morphological kidney disease
* Previous need of chronic RRT
* Prior participation in the study
* Need of extracorporeal membrane oxygenation (ECMO) or other heart assist device

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ICU, Aarhus University Hospital who are treated with dialysis as CRRT and planned to undergo dialysis weaning as determined their attending ICU physician.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Dialysis weaning | 7 days
  If discontinuation of Dialysis is successful or not. Successful dialysis weaning is defined as no renal replacement therapy (RRT) required within the first 7 days after stopping continuous renal replacement therapy (CRRT) and non-successful weaning as the need for RRT within the first 7 days.

SECONDARY OUTCOMES:
Renal Doppler arterial Resistive Index (RI) | Measured at the beginning of weaning and after 6 hours.
  Measured in the interlobar vessels
Renal Doppler Renal Venous Stasis Index (RVSI) | Measured at the beginning of weaning and after 6 hours.
  Measured in the interlobar vessels
Renal Doppler Venous Impedance Index (VII) | Measured at the beginning of weaning and after 6 hours.
  Measured in the interlobar vessels
Portal vein Doppler Pulsatility Fraction PF) | Measured at the beginning of weaning and after 6 hours.
  Measured in the interlobar vessels
Urine Output | 4 days
Urine Creatinine Clearance | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Peter Juhl-Olsen, MD, PhD, Study Chair — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Department of Anaesthesiology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No